CLINICAL TRIAL: NCT05379140
Title: Using Therapeutic Chinese Massage to Treat Peripheral Neuropathy in People With Human Immunodeficiency Virus: A Randomized Control Trial Pilot Study.
Brief Title: Use Therapeutic Chinese Massage to Treat Peripheral Neuropathy in People With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston Downtown (Other)
Responsible Party: Principal Investigator, Song Ge, Assistant Professor, University of Houston Downtown
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPHS #44-21
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Therapeutic Chinese Massage Group (Experimental): Participants in the therapeutic Chinese massage group received three weekly 25-minute therapeutic Chinese massage sessions. The intervention included acupressure to points along the distal lower extremity acupuncture points of the Gall Bladder Channel (GB 40 and then 34). Further Chinese Massage incorporates kneading, rolling, movement of the ankle, rotating, pulling, and scrubbing to the lower extremity.
  Interventions: Behavioral: Three Weekly Therapeutic Chinese Massage Sessions
- The Placebo Massage Group (Placebo Comparator): The placebo massage group received three weekly 25-minute placebo massage that included gentle rubbing to the foot and toes without point stimulation or other techniques of Chinese Massage. The control group had the opportunity to receive the treatment after the study was completed.
  Interventions: Behavioral: Three Weekly Placebo Massage Sessions

INTERVENTIONS:
Behavioral: Three Weekly Therapeutic Chinese Massage Sessions — Participants in the therapeutic Chinese massage group received three weekly 25-minute therapeutic Chinese massage sessions. The intervention included acupressure to points along the distal lower extremity acupuncture points of the Gall Bladder Channel (GB 40 and then 34). Further Chinese Massage incorporates kneading, rolling, movement of the ankle, rotating, pulling, and scrubbing to the lower extremity.
  Arms: The Therapeutic Chinese Massage Group
Behavioral: Three Weekly Placebo Massage Sessions — The placebo massage group received three weekly 25-minute placebo massage that included gentle rubbing to the foot and toes without point stimulation or other techniques of Chinese Massage. The control group had the opportunity to receive the treatment after the study was completed.
  Arms: The Placebo Massage Group

SUMMARY:
Background: Peripheral neuropathy (PN) occurs in half of the people with human immunodeficiency virus (PHIV). Currently, there is no Food and Drug Administration-approved treatment for HIV-related PN. Only half of PHIV who take medications report a significant reduction in pain. Therapeutic Chinese Massage, structured palpations or movements of soft tissues of the body, is a promising non-harmful, and non-costly intervention that can potentially alleviate or even treat PN but relevant research is limited.

Method: Investigators conducted a single centered, two-arm, single-blinded randomized controlled trial pilot study to examine if a series of three weekly 25-minute therapeutic Chinese massage sessions by a therapist of therapeutic Chinese massage, compared with placebo massage, could reduce PN-related pain and improve lower extremity functioning in PHIV. Twenty PHIV were recruited from the AIDS Foundation Houston, Inc in Texas. Pain, lower extremity functioning, and health-related quality of life were assessed for both groups prior to and post-massage.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of HIV and peripheral neuropathy have self-reported PN-related pain in lower extremity are not taking any kind of medications to alleviate PN symptoms age at least 18 years old not pregnant or lactating

Exclusion Criteria:

have received any kind of massage in the past three months Can not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of this study design | through study completion, an average of one year
  recruitment and completion rates, patient safety, and treatment adherence and compliance

SECONDARY OUTCOMES:
Change in Peripheral neuropathy related pain at the third visit | Through study completion, an average of one year
  It will be measured by the Numeric Pain Scale
Change in health related quality of life at the third visit | Through study completion, an average of one year
  It will be measured by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36)
Change in lower extremity functioning at the third visit | Through study completion, an average of one year
  It will be measured by the Lower Extremity Functioning Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston-Downtown, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ge S, Dune L, Liu M, Fu G, Ma H, Hu J, Lin X, Li J. Feasibility of therapeutic Chinese massage (tui na) for peripheral neuropathy among people with human immunodeficiency virus: findings of a pilot randomized controlled trial. Front Neurol. 2023 Dec 1;14:1148150. doi: 10.3389/fneur.2023.1148150. eCollection 2023. PMID 38107641